CLINICAL TRIAL: NCT02568319
Title: A Phase 2 Randomized, Placebo-Controlled, Double-Blind Study to Evaluate the Safety and Efficacy of LIPO-202 for the Reduction of Central Abdominal Bulging in a Defined Special Population - Obese Subjects (BMI > or Equal to 30 kg/m2)
Brief Title: Safety and Efficacy Study of LIPO-202 for the Reduction of Central Abdominal Bulging in Obese Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neothetics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LIPO-202-CL-21
Record Dates: First submitted 2015-10-02; First posted 2015-10-05 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-10

CONDITIONS: Central Abdominal Bulging
MeSH Terms: interventions — Salmeterol Xinafoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LIPO-202 (Experimental): Experimental arm
  Interventions: Drug: LIPO-202
- Placebo (Placebo Comparator): Placebo comparator
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LIPO-202
  Other Names: Salmeterol
  Arms: LIPO-202
Drug: Placebo
  Other Names: Placebo for LIPO-202
  Arms: Placebo

SUMMARY:
This is a multi-center, randomized, placebo-controlled, double-blind study evaluating the safety and efficacy of LIPO-202 for the reduction of central abdominal bulging in obese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or non-pregnant female subjects
* Capable of providing written consent
* BMI > 30 kg/m2 but < 40 kg/m2
* Stable diet and exercise routine
* At least "Slightly Dissatisfied" with their abdominal bulging on the Abdominal Contour Questionnaire (ACQ)

Exclusion Criteria:

* BMI > 40 kg/m2
* Have had any treatment of the fat around your abdomen, including surgical procedures (tummy tuck, liposuction), injections for fat loss or treatments with devices to reduce fat in your abdomen.
* Plan on starting a weight loss or exercise program during the study
* Known hypersensitivity to study drugs
* Have any medical condition that might complicate study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-09; Primary Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Safety as measured by physical examination, adverse events, vital signs, and laboratory tests. | 9 weeks
  Physical examination, adverse events, vital signs, and laboratory tests.

SECONDARY OUTCOMES:
Change in waist circumference. | 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Maria Feldman, Study Director — Neothetics, Inc
Locations (6):
- United States (6):
  - Diagnamics, Inc., Encinitas, California
  - Ablon Skin Institute and Research Center, Manhattan Beach, California
  - The Center for Clinical & Cosmetic Research, Aventura, Florida
  - Skin Research Institute, Coral Gables, Florida
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - Charlottesville Medical Research Center, Charlottesville, Virginia